CLINICAL TRIAL: NCT04265352
Title: Postnatal Managemant of Prenetal Cardiac Echogenic Foci in Hillel Yaffe
Brief Title: Postnatal Managemant of Prenetal Cardiac Echogenic Foci in Hillel Yaffe Medical Center
Status: Completed | Type: Observational
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Principal Investigator, Erez Nadir, MD, Principal investigator, Hillel Yaffe Medical Center
Other Study IDs: 0140-19-HYMC
Record Dates: First submitted 2020-01-08; First posted 2020-02-11 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Prenatal Diagnosis
Keywords: cardiac echogenic focus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prenetal cardiac echogenic focus: Newborn infants who had prenatal cardiac echogenic focus
  Interventions: Other: No intervension

INTERVENTIONS:
Other: No intervension — There is intervention at all.

SUMMARY:
Cardiac echogenic foci are common finding on prenatal follow-up. At hillel Yaffe medical center a post natal echography is performed to all newborns with prenatal cardiac echogenic foci. Reviewing the data collected until now may reduce the need for poist natal echography.

DETAILED DESCRIPTION:
Cardiac echogenic foci are common finding on prenatal follow-up. At hillel Yaffe medical center a post natal echography is performed to all newborns with prenatal cardiac echogenic foci. The investigator will review all echographies performed in the last ten years. Reviewing the data collected until now may reduce the need for poist natal echography.

ELIGIBILITY:
Inclusion Criteria:

* Newborns who had a cardiac echogenic focus during prenatal pollow-up.

Exclusion Criteria:

* Newborns who did not had postnatal echocardiography due to technical reasons.

Max Age: 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Newborn infants at hillle Yaffe medical center during 10 years: 2010-2019
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Any sonographic cardiac pathologic finding exists | 2 weeks
  Any sonographic cardiac pathologic finding exists, as defined by the cardiologist who performs the postnatal echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: Erez Nadir, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe medical center, Hadera, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No
Will not be shared

REFERENCES:
- [Background] Shakoor S, Ismail H, Munim S. Intracardiac echogenic focus and fetal outcome - review of cases from a tertiary care centre in Karachi, Pakistan. J Matern Fetal Neonatal Med. 2013 Jan;26(1):2-4. doi: 10.3109/14767058.2012.703724. Epub 2012 Jul 13. PMID 22708618